CLINICAL TRIAL: NCT04187391
Title: The Effects of a Multimodal Approach for the Treatment of Primary Progressive Aphasia
Brief Title: The Effects of a Multimodal Approach for the Treatment of PPA
Acronym: ACROSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Collaborators: Asst Degli Spedali Civili Di Brescia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GR 2018 12365105
Record Dates: First submitted 2019-11-29; First posted 2019-12-05 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Primary Progressive Aphasia
MeSH Terms: conditions — Aphasia, Primary Progressive | interventions — Language Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active tDCS plus individual language training (Experimental): Active tDCS plus individual language training
  Interventions: Device: Active tDCS; Behavioral: Language training
- placebo tDCS plus individual language training (Active Comparator): placebo tDCS plus individual language training
  Interventions: Device: Placebo tDCS; Behavioral: Language training
- Active tDCS plus unstructured cognitive stimulation (Active Comparator): Active tDCS plus unstructured cognitive stimulation
  Interventions: Device: Active tDCS; Behavioral: Unstructured cognitive training

INTERVENTIONS:
Device: Active tDCS — Active tDCS anode is applied over the left DLPFC with the cathode over the right supraorbital region.
  Arms: Active tDCS plus individual language training; Active tDCS plus unstructured cognitive stimulation
Device: Placebo tDCS — Placebo tDCS is applied but the current is turned off 10 seconds after the beginning and turned on for the last 10 seconds of the stimulation period.
  Arms: placebo tDCS plus individual language training
Behavioral: Language training — patients receive language training
  Arms: Active tDCS plus individual language training; placebo tDCS plus individual language training
Behavioral: Unstructured cognitive training — patients receive unstructured cognitive training.
  Arms: Active tDCS plus unstructured cognitive stimulation

SUMMARY:
Primary Progressive Aphasia (PPA) is an untreatable neurodegenerative disorder that disrupts language functions. Available therapies are mainly symptomatic and recently attention has been gained by new techniques that allow for noninvasive brain stimulation such as transcranial direct current stimulation (tDCS). The primary objective of this study is to evaluate whether the application of Active tDCS (anode over the left dorsolateral prefrontal cortex- DLPFC with the cathode over the right supraorbital region) to the scalp during individualized language training, would improve naming abilities in the agrammatic variant of PPA (avPPA) more than use of one methodology alone. The effect of treatment on the clinical symptoms will be related to changes in brain activity (Magnetic Resonance Imaging, MRI and Functional near-infrared spectroscopy fNIRS) and in biological markers, using a multimodal approach. Finally, we will assess the long-term effects of this approach.

DETAILED DESCRIPTION:
45 patients with avPPA, will be recruited from IRCCS Istituto Centro San Giovanni di Dio Brescia, Italy and ASST Spedali Civili Brescia, Italy .

Inclusion criteria will be a diagnosis avPPA according to the current clinical criteria (Gorno-Tempini et al., 2011) and a FTD Clinical Dementia Rating score >0.5 and <2. Exclusion criteria will be the presence of any medical or psychiatric illness that could interfere in completing assessments and the presence of any medical condition that represents a contraindication to tDCS. All the patients will undergo five consecutive days a week for two weeks of treatment sessions:

15 patients will receive Active tDCS over DLPFC while performing a language training; 15 patients will receive placebo tDCS during language training; 15 patients will receive Active tDCS over DLPFC during unstructured cognitive training.

Two trained neuropsychologists will administer the neuropsychological testing in two sessions. At baseline (T0), post-treatment (T1) and 3-months (T2) follow-up assessments were conducted by the same assessor. Blood sample withdrawal at baseline (T0) and after the DLPFC-tDCS intervention (T1) will be assessed.

To elucidate the mechanisms underlying tDCS effects, structural imaging, functional connectivity (fMRI) alterations and concentration changes of hemoglobin (fNIRS) will be collected off-line. Each avPPA patient will undergo an MRI scan at the ASST Spedali Civili Brescia, Italy at T0 and T1 and a fNIRS acquisition at the IRCCS Istituto Centro San Giovanni di Dio Brescia, Italy at T0, T1 and T2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis avPPA according to the current clinical criteria (Gorno-Tempini et al., 2011)
* FTD Clinical Dementia Rating (FTD-CDR) score >0.5 and <2

Exclusion Criteria:

* Presence of any medical or psychiatric illness that could interfere in completing assessments
* Presence of any medical condition that represents a contraindication to tDCS.

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in naming test scores on Picture Naming Task | Baseline up to 2 weeks and 3 months
  Picture Naming Task: percentage of correct responses (0-100)

SECONDARY OUTCOMES:
Change in quality of life on Stroke and Aphasia Quality of Life | Baseline up to 2 weeks and 3 months
  Stroke and Aphasia Quality of Life (0-5; higher scores=better quality of life)
Change in dementia severity on Frontotemporal Dementia-modified Clinical Dementia Rating Scale | Baseline up to 2 weeks and 3 months
  Frontotemporal Dementia-modified Clinical Dementia Rating Scale (0-3; higher scores=greater dementia severity)
Change in cognitive impairment on Mini Mental State Examination | Baseline up to 2 weeks and 3 months
  Mini Mental State Examination (0-30; higher scores=better cognitive abilities)
Change in verbal long term memory on Story Recall | Baseline up to 2 weeks and 3 months
  Story Recall (0-28; higher scores=better memory abilities)
Change in nonverbal long term memory on Rey-Osterrieth Complex Figure-Recall | Baseline up to 2 weeks and 3 months
  Rey-Osterrieth Complex Figure-Recall (0-36; higher scores=better abilities)
Change in attentional abilities on Trial Making Test | Baseline up to 2 weeks and 3 months
  Trial Making Test (milliseconds; higher scores=worse abilities)
Change in constructional praxia on Rey-Osterrieth Complex Figure-Copy | Baseline up to 2 weeks and 3 months
  Rey-Osterrieth Complex Figure-Copy (0-36; higher scores=better abilities)
Change in fluency abilities on Verbal Fluency (semantic and phonemic) | Baseline up to 2 weeks and 3 months
  Verbal Fluency (semantic and phonemic) Test (higher scores=better abilities)
Change in aphasia severity on Screening for Neurodegenerative Aphasia | Baseline up to 2 weeks and 3 months
  Screening for Neurodegenerative Aphasia Battery (higher scores=better abilities)
Change in naming on naming subtest from Aachener Aphasie Test | Baseline up to 2 weeks and 3 months
  naming subtest from Aachener Aphasie Test (0-120; higher scores=better abilities)
Change in language impairment on Mini Language State Examination | Baseline up to 2 weeks and 3 months
  Mini Language State Examination Battery (higher scores=better abilities)
Change in molecular biomarkers on neurogranin | Baseline up to 2 weeks
  neurogranin
Change in imaging biomarkers on fMRI and fNIRS | Baseline up to 2 weeks
  fMRI and fNIRS

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Manenti, PhD, Principal Investigator — IRCCS Istituto Centro San Giovanni di Dio- Fatebenefratelli
Locations (1):
- IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: Undecided